CLINICAL TRIAL: NCT05987410
Title: EffectiVenEss of a Rehabilitation Treatment With Nordic Walking in obEse or oveRweight Diabetic patiEnts With Cardiovascular Disease. The VENERE Study
Brief Title: EffectiVenEss of a Rehabilitation Treatment With Nordic Walking in obEse or oveRweight Patients
Acronym: VENERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Nuccia Morici, MD, Ph.D., Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 27/2023/CE_FdG/FC/SA
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases; Diabete Type 2; Overweight and Obesity
Keywords: Nordic Walking (NW); cardiovascular disease; diabetes Type II; overweight; obesity; Six Minute Walking Test (6MWT); adherence; rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — Nordic Walking

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized controlled intervention study with three parallel arms (NW=Nordic Walking, SR=standard rehabilitation and CG=control group), open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nordic Walking (NW) (Experimental): Nordic walking is a form of physical activity that originated in Finland and has gained popularity worldwide. It involves walking with the use of specially designed poles that resemble ski poles. This activity engages both the upper and lower body, making it a full-body workout. In summary, Nordic walking offers several benefits for cardiovascular individuals with Type II diabetes and those who are obese or overweight. These benefits include improved heart and lung function, better blood glucose control, weight management, low joint impact, muscle strengthening, improved balance and posture, and social engagement. However, it is important to consult with a healthcare provider before starting any new exercise program to ensure it is safe and suitable for individual health conditions and goals. Regular monitoring and adjustments by healthcare professionals can help optimize the benefits and ensure ongoing progress.
  Interventions: Other: Nordic Walking (NW)
- Standard Rehabilitation (SR) (Active Comparator): A standard rehabilitation program for cardiovascular individuals with Type II diabetes and obesity/overweight typically involves a combination of cardiovascular exercise, strength training, and education on lifestyle modifications. The program is prescribed by a cardiologist and supervised by physiotherapists or exercise specialists. It includes an initial assessment to determine exercise parameters, cardiovascular exercise to improve heart function and manage blood glucose levels, strength training to increase muscle mass and aid in weight management, education on nutrition and lifestyle modifications, and progress tracking and monitoring to optimize outcomes. These programs provide benefits such as improved cardiovascular fitness, better blood glucose control, weight management, enhanced muscle strength, and overall well-being.
  Interventions: Other: Standard Rehabilitation (SR)
- Control Group (CG) (Other): Cardiological counseling for cardiovascular individuals with Type II diabetes and obesity/overweight often includes recommendations for unsupervised aerobic physical activity. This type of counseling typically involves a cardiologist providing guidelines and recommendations for safe and effective exercise routines. In summary, it involves an initial assessment to determine exercise capacity and precautions. The cardiologist prescribes specific guidelines for unsupervised aerobic physical activity, including the type, frequency, intensity, and duration of exercise sessions. Safety considerations are provided. The benefits of unsupervised aerobic physical activity include improved cardiovascular health, enhanced blood glucose control, weight management, psychological well-being, and increased energy and stamina.
  Interventions: Other: Cardiological Counselling (CC)

INTERVENTIONS:
Other: Nordic Walking (NW) — The experimental group will carry out NW sessions three times a week for 12 weeks, supervised by a NW instructor and under the control of a cardiologist. The duration of each NW session will initially be 90 minutes: 10 minutes of warm-up, 60 of NW, and 15 minutes of cool-down. The intensity of the course will be gradually increased each week, starting at 70 to 85% of the heart rate (HR) reserve. It will also receive indications relating to a balanced diet plan which proposes a moderate (300-400 KCal) daily caloric restriction concerning the usual caloric expenditure, estimated based on initial body composition measurements.
  Arms: Nordic Walking (NW)
Other: Standard Rehabilitation (SR) — The second group will follow a standard rehabilitation program with an initial cardiological prescription and supervised by physiotherapists, carried out 5 days a week with sessions lasting 40 minutes, including 5 minutes of warm-up up), 30 min of aerobic physical activity on a conveyor belt or cycle ergometer and 5 minutes of cooling down (cool down). The intensity of your aerobic activity will gradually increase each week, starting at 70 to 85% of HR reserve. It will also receive indications relating to a balanced diet plan which proposes a moderate (300-400 KCal) daily caloric restriction concerning the usual caloric expenditure, estimated based on initial body composition measurements.
  Arms: Standard Rehabilitation (SR)
Other: Cardiological Counselling (CC) — The third group of participants will receive cardiological counselling with indications of unsupervised aerobic physical activity. The group will also receive indications relating to a balanced diet plan which proposes a moderate (300-400 KCal) daily caloric restriction concerning the usual caloric expenditure, estimated based on initial body composition measurements.
  Arms: Control Group (CG)

SUMMARY:
Nordic Walking (NW) is a biomechanically correct walking technique that originated in Finland in the 1930s as an off-season training method for cross-country skiers. In the NW, the use of special sticks is combined with "conventional" walking: this involves a greater caloric expenditure, with an energy consumption higher by 20-30% compared to walking without sticks, and also toning of the upper part of the body, in particular triceps, shoulders and back, and the involvement of about 90% of the body's muscles, while maintaining a reduced load on ligaments and joints (Baek & Ha, 2021). The NW acts simultaneously and effectively on different components of fitness: coordination, endurance, strength, and mobility. It does not require sudden accelerations and is based on a technique that is easy to learn (with the help of an instructor), especially as regards maintaining correct posture. Finally, in addition to the cardiovascular benefits, NW has also been shown to effectively reduce the risk of falls in the elderly. The study is a single-center, randomized controlled trial (RCT), with a three-parallel-arm design, open-label. The primary objective is to evaluate the efficacy (in terms of cardiovascular performance), safety, and adherence (in terms of dropout rate) to the exercise prescription after 6 and 12 months follow-up of a 3-month NW intervention compared with standard rehabilitation training (SR, 3 months) in obese/overweight diabetic patients with cardiovascular (CV) complications. The study will enroll in parallel a control group that can access only generic cardiological counseling with a prescription for unsupervised home exercise.

ELIGIBILITY:
Inclusion Criteria:

- overweight [Body Mass Index (BMI) ≥ 27 kg/m2] or obese (BMI ≥30 kg/m2) adult patients with diabetes mellitus and with a recent cardiovascular event and/or coronary revascularization in the previous three months

Exclusion Criteria:

* inability to walk independently and constantly;
* acute joint or spine pathologies that make movement impossible;
* the presence of dementia as approved by consultation of the patient's medical record and/or administration of the Montreal Cognitive Assessment (MOCA) test ≤ 15.5 (Nasreddine et al., 2005);
* chemotherapy 6 months before surgery;
* advanced renal failure;
* acute cardiovascular event < 3 months (unstable angina, AMI with FE <40%, arrhythmias, valvular disease, intracerebral/subdural haemorrhage, uncontrolled AI);
* home oxygen therapy and Non-Invasive Ventilation (NIV) [excluding Continuous Positive Airway Pressure (CPAP)].

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walking Test (6MWT) distance in meters | An average of 6 months
  Assess distance in meters, determined by the Six Minute Walking Test (6MWT) in the Nordic Walking (NW) group compared to the Standard Rehabilitation (SR) and Control (CG) Groups at baseline (T0), the end of the rehabilitation treatment (T1), and after 3 months of observation (T2)

SECONDARY OUTCOMES:
Adherence | Through intervention completion, an average of 3 months
  Monitoring of adherence to the intervention considering the number of sessions of the treatment [Nordic Walking (NW); Standard Rehabilitation (SR) or Control Group (CG) intervention] attended during the 3 months.
Anxiety | An average of 6 months
  To verify the effectiveness of the interventions in reducing the levels of anxiety as detected by The Generalized Anxiety Disorder Scale (GAD-7) in the Nordic Walking (NW) group compared to the Standard Rehabilitation (SR) and Control (CG) Groups at baseline (T0), the end of the rehabilitation treatment (T1), and after 3 months of observation (T2). The following cut-offs correlate with level of anxiety severity: Score 0-4: Minimal Anxiety; Score 5-9: Mild Anxiety; Score 10-14: Moderate Anxiety; Score greater than 15: Severe Anxiety (Spitzer et al., 2006).
Depression | An average of 6 months
  To verify the effectiveness of the interventions in reducing the levels of depression as detected by The Patient Health Questionnaire-9 (PHQ-9) in the Nordic Walking (NW) group compared to the Standard Rehabilitation (SR) and Control (CG) Groups at baseline (T0), the end of the rehabilitation treatment (T1), and after 3 months of observation (T2). Regarding severity, PHQ-9 comprises five categories, where a cut-off point of 0-4 indicates no depressive symptoms, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately-severe depressive symptoms, and 20-27 severe depressive symptoms (Kroenke and Spitzer, 2002).
The Short Form Health Survey 12 (SF-12) | An average of 12 months
  To verify the effectiveness of the interventions in improving the levels of Quality of Life detected thanks to The Short Form Health Survey 12 (SF-12) (Ware et al., 2000) in the Nordic Walking (NW) group compared to the Standard Rehabilitation (SR) and Control (CG) Groups at baseline (T0), the end of the rehabilitation treatment (T1), after 3 months of observation (T2), 12 months (T3).
Variation in Body Mass Index (BMI) | An average of 12 months
  To verify the effectiveness of the interventions in improving the Body Mass Index (BMI) in the Nordic Walking (NW) group compared to the Standard Rehabilitation (SR) and Control (CG) Groups at baseline (T0), the end of the rehabilitation treatment (T1), after 3 months of observation (T2), 12 months (T3).
  An improvement of at least 10% in BMI is considered significant.
Peak Oxygen Uptake (VO2) | An average of 6 months
  Assess increasing in Peak Oxygen Uptake (VO2) in the Nordic Walking (NW) group compared to the Standard Rehabilitation (SR) and Control (CG) Groups group at baseline (T0), the end of the rehabilitation treatment (T1), and after 3 months of observation (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Torri, MD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohammad NS, Nazli R, Zafar H, Fatima S. Effects of lipid based Multiple Micronutrients Supplement on the birth outcome of underweight pre-eclamptic women: A randomized clinical trial. Pak J Med Sci. 2022 Jan-Feb;38(1):219-226. doi: 10.12669/pjms.38.1.4396. PMID 35035429
- [Background] Conroy DE, Maher JP, Elavsky S, Hyde AL, Doerksen SE. Sedentary behavior as a daily process regulated by habits and intentions. Health Psychol. 2013 Nov;32(11):1149-57. doi: 10.1037/a0031629. Epub 2013 Mar 11. PMID 23477579
- [Background] Despres JP, Carpentier AC, Tchernof A, Neeland IJ, Poirier P. Management of Obesity in Cardiovascular Practice: JACC Focus Seminar. J Am Coll Cardiol. 2021 Aug 3;78(5):513-531. doi: 10.1016/j.jacc.2021.05.035. PMID 34325840
- [Background] Elavsky S, McAuley E. Physical activity and mental health outcomes during menopause: a randomized controlled trial. Ann Behav Med. 2007 Apr;33(2):132-42. doi: 10.1007/BF02879894. PMID 17447865
- [Background] Gholami M, Larijani B, Zahedi Z, Mahmoudian F, Bahrami S, Omran SP, Saadatian Z, Hasani-Ranjbar S, Taslimi R, Bastami M, Amoli MM. Inflammation related miRNAs as an important player between obesity and cancers. J Diabetes Metab Disord. 2019 Nov 26;18(2):675-692. doi: 10.1007/s40200-019-00459-2. eCollection 2019 Dec. PMID 31890692
- [Background] Henning RJ. Obesity and obesity-induced inflammatory disease contribute to atherosclerosis: a review of the pathophysiology and treatment of obesity. Am J Cardiovasc Dis. 2021 Aug 15;11(4):504-529. eCollection 2021. PMID 34548951
- [Background] La Sala L, Pontiroli AE. Prevention of Diabetes and Cardiovascular Disease in Obesity. Int J Mol Sci. 2020 Oct 31;21(21):8178. doi: 10.3390/ijms21218178. PMID 33142938
- [Background] Ipp E, Genter P, Childress K. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2017 Mar 2;376(9):890-1. doi: 10.1056/NEJMc1615712. No abstract available. PMID 28252263
- [Background] Baek S, Ha Y, Park HW. Accuracy of Wearable Devices for Measuring Heart Rate During Conventional and Nordic Walking. PM R. 2021 Apr;13(4):379-386. doi: 10.1002/pmrj.12424. Epub 2020 Jul 17. PMID 32449291
- [Background] Graffigna G, Barello S, Bonanomi A, Lozza E, Hibbard J. Measuring patient activation in Italy: Translation, adaptation and validation of the Italian version of the patient activation measure 13 (PAM13-I). BMC Med Inform Decis Mak. 2015 Dec 23;15:109. doi: 10.1186/s12911-015-0232-9. PMID 26699852
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Derived] Torri A, Volpato E, Merati G, Milani M, Toccafondi A, Formenti D, La Rosa F, Agostini S, Agliardi C, Oreni L, Sacco A, Rescaldani M, Lucreziotti S, Giglio A, Ferrante G, Barbaro M, Montalto C, Buratti S, Morici N. The VENERE Study: EffectiVenEss of a Rehabilitation Treatment With Nordic Walking in ObEse or OveRweight Diabetic PatiEnts With Cardiovascular Disease. CJC Open. 2024 Jan 16;6(5):735-744. doi: 10.1016/j.cjco.2024.01.002. eCollection 2024 May. PMID 38846444